CLINICAL TRIAL: NCT00814177
Title: Management of Prothrombin Times Outside the Therapeutic Range in Patients on Warfarin and With Otherwise Stable Levels
Brief Title: Prothrombin Times Outside the Therapeutic Range in Otherwise Stable Patients
Acronym: FORESPEAK-0
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Sam Schulman, Professor, MD, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRC060425
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Results first posted 2009-11-25 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism; Ischemic Stroke; Myocardial Infarction
Keywords: warfarin; dosing; prothrombin time; Heart valve prosthesis
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism; Ischemic Stroke; Myocardial Infarction | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No change (Experimental): Intervention Drug warfarin no change in the dose is performed
  Interventions: Drug: warfarin
- Change (Active Comparator): Intervention Drug Warfarin One dose increased if subtherapeutic level; one dose deleted or reduced if supratherapeutic level
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: warfarin — No change: Continue without any change in spite of prothrombin time outside the therapeutic range.
  Other Names: Coumadin
  Arms: No change
Drug: warfarin — Change: Increase one dose in case prothrombin time is below the therapeutic range; delete or reduce one dose in case prothrombin time is above the therapeutic range.
  Other Names: Coumadin
  Arms: Change

SUMMARY:
Warfarin is very effective for the prevention of blood clots (thrombosis). A test of coagulation, the prothrombin time (PT) is used to monitor the effect. The PT response to warfarin can fluctuate as a result of interactions with a large number of other drugs, food or herbal agents as well as for no apparent reason. Thus, frequent monitoring of the PT and dose adjustments according to the results are required. One third of our patients remain on the same maintenance dose over 6 months. However, also these patients sometimes have a PT result moderately outside the therapeutic range without any obvious explanation. Too short PTs may be due to missed dose(s) or more dark green vegetables in the diet. Too long PTs may be due to a course of antibiotic therapy or less dark green vegetables. Laboratory errors may also occur and can cause deviations in any direction. Most likely, unnoticed fluctuations in the PT occur as well between the time points of monitoring.

There are no guidelines on how to manage the treatment in this situation but there are some typical "behaviours".

Behavior A: Some physicians simply let the patient continue with the same dose. "It is extremely unlikely that the very temporary dose adjustment has any effect on the PT result 4 weeks later and this is a "cosmetic procedure"." Behavior B: Others recommend the patients to take ½ - 1 additional dose in case of short PT and to skip a dose or take half dose in case of long PT, and thereafter to continue with the usual dose. "The investigators need to quickly correct the temporary aberration in order to avoid thrombotic or bleeding complications the next few days.

This may seem like an issue of no importance. The investigators are however performing a series of studies to evaluate if these stable patients can be managed with blood tests less often than every 4 weeks. For that purpose it is important to know how often and why aberrant results occur, the implication and to what extent they can be ignored.

The investigators hypothesis is that in patients with very stable PT-results and unchanged dose for 3 months, should continue with exactly the same maintenance dose, even when the result unexpectedly is slightly above or below the therapeutic range. The investigators believe that most of these occasional PT-results outside the therapeutic range are due to laboratory errors, perhaps missed doses by the patient or temporary change in diet or medications.

DETAILED DESCRIPTION:
Setting:

Thrombosis Service at HHS - General Hospital. This center monitors the warfarin treatment for 1300 patients in the region. These patient regularly go to a laboratory where they live. Test results (INR-results) are faxed to the Thrombosis Service, which calls the patient the same day to inform them of the results, how to continue dosing the warfarin and when to go for the following blood test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on long-term warfarin (for prophylaxis of arterial embolism in patients with atrial fibrillation or mechanical heart valve replacement, or secondary prophylaxis after VTE) with a target INR of 2.0-3.0 or 2.5-3.5,
2. Anticoagulant therapy managed by the clinic (HHS - General Hospital) for at least 3 months prior to enrolment, and
3. Maintenance dose of warfarin unchanged for the previous 3 months or longer.
4. The INR result is outside the therapeutic range as follows:

For those with target 2.0-3.0: Either an INR of 1.5-1.9 or an INR of 3.1-4.4. For those with target 2.5-3.5: Either an INR of 1.5-2.4 or an INR of 3.6-4.4.

Exclusion Criteria:

1. Age <18 years,
2. Long-term (>1 week) change in any other medication
3. Long-term (>1 week) change in diet, especially regarding green vegetables.
4. Attending physician believes the patient is not suitable for the study (e.g. psychiatric disorder, history of non-compliance),
5. Failure to obtain telephone consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schulman, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Thrombosis Service, HHS-General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Schulman S, Melinyshyn A, Ennis D, Rudd-Scott L. Single-dose adjustment versus no adjustment of warfarin in stably anticoagulated patients with an occasional international normalized ratio (INR) out of range. Thromb Res. 2010 May;125(5):393-7. doi: 10.1016/j.thromres.2009.07.006. Epub 2009 Jul 29. PMID 19640572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 160 patients were randomized at a single center during the period July 2006 - August 2008
Pre-assignment Details: The study was planned for the sample size of 326 but due to competing studies, testing new dosing algorithms, the inclusion rate was much lower than expected.
Period: Overall Study
Arm/Group | No Change | Change
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Change | Change | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 33 | 54
  >=65 years | 59 | 47 | 106
Age Continuous [Mean (Standard Deviation); unit: years] | 69.6 (11.4) | 67.1 (13.8) | 68.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 49 | 46 | 95
Region of Enrollment [Number; unit: participants]
  Canada | 80 | 80 | 160

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Prothrombin Time Results Within the Therapeutic Range After 2 Weeks
Description: The number of patients with "follow-up INRs" within the therapeutic range was compared for patients with a single dose skipped/reduced/added versus patients with no change of dose.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | No Change | Change
Number analyzed (Participants) | 80 | 80
participants | 48 | 45

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | No Change | Change
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 2/80 | 1/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Change (N=80) | Change (N=80)
ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — triggered by implanted defibrillator malfunction
food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
bleeding from penis (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No